CLINICAL TRIAL: NCT05461794
Title: Phase 2, Randomized, Open-Label Study to Investigate the Efficacy and Safety of Sitravatinib in Combination With Tislelizumab in Patients With Locally Advanced Unresectable or Metastatic Esophageal Squamous Cell Carcinoma That Progressed on or After Anti-PD-(L)1 Antibody Therapy
Brief Title: Study To Investigate the Efficacy and Safety of Sitravatinib in Combination With Tislelizumab in Participants With Esophageal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to modification of company strategy.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-Sitravatinib-203; CTR20222088 (Other: ChinaDrugTrials)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sitravatinib; tislelizumab; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Tislelizumab + Sitravatinib (Experimental): Sitravatinib administered orally and tislelizumab administered intravenously
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab
- Arm B: Sitravatinib (Experimental): Sitravatinib administered orally
  Interventions: Drug: Sitravatinib
- Arm C: Investigator-chosen chemotherapy (ICC) (Experimental): Investigators chose between docetaxel or irinotecan
  Interventions: Drug: Docetaxel; Drug: Irinotecan

INTERVENTIONS:
Drug: Sitravatinib — 100 mg orally once daily
  Other Names: BGB-9468
  Arms: Arm A: Tislelizumab + Sitravatinib; Arm B: Sitravatinib
Drug: Tislelizumab — 200 mg intravenously once every 3 weeks
  Other Names: BGB-A317
  Arms: Arm A: Tislelizumab + Sitravatinib
Drug: Docetaxel — 75 milligrams per square meter of body surface area (mg/m2) intravenously on Day 1 of every 21-day cycle
  Arms: Arm C: Investigator-chosen chemotherapy (ICC)
Drug: Irinotecan — 125 mg/m2 intravenously on Days 1 and 8 of every 21-day cycle
  Arms: Arm C: Investigator-chosen chemotherapy (ICC)

SUMMARY:
The study aimed to evaluate the efficacy and safety of sitravatinib in combination with tislelizumab as a second- or third-line treatment for participants with locally advanced, unresectable, or metastatic esophageal squamous cell carcinoma (ESCC) who experienced disease progression following prior systemic chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced unresectable or metastatic ESCC, not amenable to treatment with curative intent
2. At least 1 measurable lesion as defined per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as determined by local site investigator/radiology assessment ≤ 28 days before randomization Note: Lesions that had been previously irradiated were considered evaluable provided
3. Eastern Cooperative Oncology Group (ECOG) score ≤ 1
4. Adequate organ function as indicated by the following laboratory values as indicated by the laboratory tests performed ≤ 7 days before randomization

Key Exclusion Criteria:

1. Have any contraindication for receiving treatment with both docetaxel and irinotecan
2. Participants with tumor located around important vascular structures as shown by imaging or the investigator determines that the tumor is likely to invade important blood vessels and may cause fatal bleeding (ie, radiologic evidence of tumors invading or abutting major blood vessels)
3. Participants with tumor that invades into organs located adjacent to the esophageal disease site (eg, aorta or respiratory tract) that has an increased risk of fistula during the study treatment period as assessed by the investigator
4. History of gastrointestinal perforation and/or fistula or aorto-esophageal fistula within 6 months before randomization
5. Have received prior anticancer agents that have same mechanism of action as sitravatinib (eg, receptor tyrosine kinases (RTKs) with a similar target profile or Vascular Endothelial Growth Factor (VEGF)/Vascular Endothelial Growth Factor Receptor-targeted (VEGFR) monoclonal antibodies)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Anhui Provincial Hospital South Brance, Hefei, Anhui
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat Sen University Cancer Center(Huangpu Campus), Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Northern Jiangsu Peoples Hospital, Yangzhou, Jiangsu
  - Ganzhou Peoples Hospital Ganzhou Hospital Affiliated to Nanchang University, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across multiple study centers in China. The first participant provided consent on October 3, 2022, and the last participant completed the study on February 26, 2024.
Pre-assignment Details: Participants were randomly assigned to one of three treatment groups in a 2:1:2 ratio. Randomization was stratified by PD-L1 expressions status (Tumor Area Positivity [TAP] score ≥ 10% versus TAP score < 10%)
Groups:
- Arm A: Tislelizumab + Sitravatinib: Sitravatinib was administered orally at a dose of 100 mg once daily, while tislelizumab was given intravenously at 200 mg once every three weeks.
- Arm B: Sitravatinib: Sitravatinib was administered orally at a dose of 100 mg once daily.
- Arm C: Investigator-chosen Chemotherapy (ICC): Investigators selected either docetaxel, administered intravenously at 75 mg/m² on Day 1 of each 21-day cycle, or irinotecan, given intravenously at 125 mg/m² on Days 1 and 8 of each 21-day cycle.
Period: Overall Study
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
Started | 39 | 19 | 38
Treated | 39 | 19 | 34
Completed | 0 | 0 | 0
Not Completed | 39 | 19 | 38
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Study Terminated By Sponsor | 18 | 13 | 16
Not completed — Death | 20 | 5 | 19

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) analysis set included all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC) | Total
Number analyzed (Participants) | 39 | 19 | 38 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (7.73) | 61.9 (7.87) | 60.4 (8.06) | 60.2 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 37 | 17 | 35 | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 39 | 19 | 38 | 96

OUTCOME MEASURES:

1. Primary Outcome: Arms A and C: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) as assessed by the investigator per the Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1.
Time Frame: Through study completion data cut-off date of February 26th, 2024 (maximum time on study was 12 months)
Population: The Intent-to-Treat (ITT) analysis set included all randomized participants; for the primary analysis of ORR only Arms A and C were included, results for Arm B are included in the secondary Outcome Measures section.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
Number analyzed (Participants) | 39 | 38
percentage of participants | 10.3 [2.9 to 24.2] | 5.3 [0.6 to 17.7]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm C: Investigator-chosen Chemotherapy (ICC); Test type: Other; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.3 to 23.9] — The crude odds ratio was estimated along with exact unconditional 95% CIs constructed by the tail method based on the score statistics
Statistical Analysis 2: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm C: Investigator-chosen Chemotherapy (ICC); Test type: Other; Risk Difference (RD) = 5.0, 95% CI 2-sided [-9.3 to 19.5] — The risk difference was estimated along with their exact unconditional 95% CIs constructed by the tail method based on the score statistics

2. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from the first occurrence of a documented objective response to the time of documented disease progression assessed by the investigator or death from any cause, whichever occurred first, in all randomized participants with documented objective responses.
Time Frame: Through study completion data cut-off date of February 26th, 2024 (maximum time on study was 12 months)
Population: ITT analysis Set. Only participants with best overall response of complete response or partial response confirmed per RECIST v1.1 were included in the analysis, and percentages were based on the number of responders
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
Number analyzed (Participants) | 4 | 4 | 2
months | 5.2 [4.4 to NA] — Not estimable due to insufficient number of participants with events | 4.6 [2.8 to NA] — Not estimable due to insufficient number of participants with events | NA [2.8 to NA] — Not estimable due to insufficient number of participants with events

3. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from randomization until the date of death due to any cause. Kaplan-Meier methodology was used to estimate the median OS.
Time Frame: Through study completion data cut-off date of February 26th, 2024 (maximum time on study was 12 months)
Population: ITT analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
Number analyzed (Participants) | 39 | 19 | 38
months | 6.1 [3.4 to 7.5] | 9.1 [6.5 to NA] — Not estimable due to insufficient number of participants with events | 5.5 [4.7 to 6.6]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm C: Investigator-chosen Chemotherapy (ICC); Test type: Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.45 to 1.61] — Hazard ratio and 95% CIs were estimated using a Cox regression model stratified by PD-L1 tumor area positivity score (>=10% versus < 10%)

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Defined as the percentage of participants whose best overall response is complete response, partial response, or stable disease, as assessed by the investigator per RECIST v1.1
Time Frame: Through study completion data cut-off date of February 26th, 2024 (maximum time on study was 12 months)
Population: ITT analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
Number analyzed (Participants) | 39 | 19 | 38
percentage of participants | 64.1 [47.2 to 78.8] | 63.2 [38.4 to 83.7] | 42.1 [26.3 to 59.2]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm C: Investigator-chosen Chemotherapy (ICC); Test type: Other; Odds Ratio (OR) = 2.5, 95% CI 2-sided [0.9 to 6.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm B: Sitravatinib; Test type: Other; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.3 to 3.7] — The odds ratio was estimated along with their exact unconditional 95% CIs constructed by the tail method based on the score statistics
Statistical Analysis 3: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm C: Investigator-chosen Chemotherapy (ICC); Test type: Other; Risk Difference (RD) = 22.0, 95% CI 2-sided [-1.5 to 43.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm B: Sitravatinib; Test type: Other; Risk Difference (RD) = 0.9, 95% CI 2-sided [-24.5 to 28.4] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Defined as the percentage of participants with a complete response, partial response, or durable stable disease (defined as stable disease for 24 weeks or longer, as assessed by the investigator per RECIST v.1.1.
Time Frame: Through study completion data cut-off date of February 26th, 2024 (maximum time on study was 12 months)
Population: ITT analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
Number analyzed (Participants) | 39 | 19 | 38
percentage of participants | 17.9 [7.5 to 33.5] | 26.3 [9.1 to 51.2] | 5.3 [0.6 to 17.7]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm C: Investigator-chosen Chemotherapy (ICC); Test type: Other; Odds Ratio (OR) = 3.9, 95% CI 2-sided [0.7 to 40.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm B: Sitravatinib; Test type: Other; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.1 to 2.9] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm C: Investigator-chosen Chemotherapy (ICC); Test type: Other; Risk Difference (RD) = 12.7, 95% CI 2-sided [-2.3 to 29.5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm B: Sitravatinib; Test type: Other; Risk Difference (RD) = -8.4, 95% CI 2-sided [-34.7 to 13.8] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the time from randomization until first documentation of disease progression as assessed by the investigator per RECIST v1.1 or death from any cause, whichever occurred first. Kaplan-Meier methodology was used to estimate the median PFS.
Time Frame: Through study completion data cut-off date of February 26th, 2024 (maximum time on study was 12 months)
Population: ITT analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
Number analyzed (Participants) | 39 | 19 | 38
months | 3.4 [2.1 to 5.6] | 5.6 [2.1 to NA] — Not estimable due to insufficient number of participants with events | 2.6 [1.5 to 3.8]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm C: Investigator-chosen Chemotherapy (ICC); Test type: Other; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.29 to 0.96] — Hazard ratio and 95% CIs were estimated using a Cox regression model stratified by the selected stratification factors PD-L1 tumor area positivity score (>=10% versus < 10%)
Statistical Analysis 2: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm B: Sitravatinib; Test type: Other; Hazard Ratio (HR) = 1.96, 95% CI 2-sided [0.79 to 4.82] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Arms A and B: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) as assessed by the investigator per RECIST v1.1. Analysis of ORR in Arm A compared to Arm B was specified as a secondary endpoint in the Protocol (please see the primary outcome measure for Arm C results)
Time Frame: Through study completion data cut-off date of February 26th, 2024 (maximum time on study was 12 months)
Population: ITT analysis set for Arms A and B
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib
Number analyzed (Participants) | 39 | 19
percentage of participants | 10.3 [2.9 to 24.2] | 21.1 [6.1 to 45.6]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Sitravatinib vs Arm B: Sitravatinib; Test type: Other; Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.1 to 2.7] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), which includes laboratory tests, and vital signs, according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Time Frame: From the first dose to 30 days after the last dose or the start of new anticancer therapy, whichever occurred first (maximum time on treatment was 8.9 months for Arm A, 7.7 months for Arm B, and 8.0 months for Arm C).
Population: The Safety Analysis Set includes all participants who received at least 1 dose of any component of study treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
Number analyzed (Participants) | 39 | 19 | 34
Participants
  TEAEs | 39 | 19 | 34
  SAEs | 22 | 6 | 15

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed through the end of study, February 26th, 2024 (maximum time on study was 12 months). Adverse events were assessed from the first dose of study drug to 30 days after the last dose or the start of new anticancer therapy, whichever occurred first (maximum time on treatment was 8.9 months for Arm A, 7.7 months for Arm B, and 8.0 months for Arm C).
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events includes all randomized participants who received ≥ 1 dose of any study treatment.
Arm/Group | Arm A: Tislelizumab + Sitravatinib | Arm B: Sitravatinib | Arm C: Investigator-chosen Chemotherapy (ICC)
All-Cause Mortality (participants affected / at risk) | 20/39 | 5/19 | 19/38
Serious Adverse Events (participants affected / at risk) | 22/39 | 6/19 | 15/34
Other Adverse Events (participants affected / at risk) | 39/39 | 19/19 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tislelizumab + Sitravatinib (N=39) | Arm B: Sitravatinib (N=19) | Arm C: Investigator-chosen Chemotherapy (ICC) (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumopericardium (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 5 (5) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tislelizumab + Sitravatinib (N=39) | Arm B: Sitravatinib (N=19) | Arm C: Investigator-chosen Chemotherapy (ICC) (N=34)
Anaemia (Blood and lymphatic system disorders) | 12 (18) | 5 (6) | 20 (23)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve calcification (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Central hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 9 (10) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 3 (4) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (11) | 1 (1) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 3 (4) | 14 (28)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 12 (14)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 10 (12)
Asthenia (General disorders) | 6 (6) | 4 (5) | 3 (3)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 4 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 2 (3)
Malaise (General disorders) | 3 (4) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (7) | 0 (0) | 5 (7)
COVID-19 (Infections and infestations) | 4 (5) | 2 (7) | 4 (8)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (22) | 6 (7) | 4 (9)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 3 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 15 (25) | 9 (11) | 2 (2)
Bilirubin conjugated increased (Investigations) | 1 (1) | 1 (2) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 1 (2) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (4) | 1 (1) | 3 (3)
Blood creatine phosphokinase MB increased (Investigations) | 6 (11) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (5) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 6 (8) | 2 (3) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 4 (4) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (3) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (2) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 1 (1) | 2 (2)
High density lipoprotein decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (4) | 0 (0) | 5 (6)
Neutrophil count decreased (Investigations) | 3 (3) | 5 (15) | 21 (48)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 9 (16) | 7 (9) | 6 (10)
Red blood cells urine positive (Investigations) | 0 (0) | 1 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 3 (3) | 1 (2) | 2 (2)
Urinary occult blood positive (Investigations) | 2 (2) | 1 (2) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 10 (11) | 7 (8) | 9 (12)
White blood cell count decreased (Investigations) | 7 (12) | 5 (15) | 24 (55)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 7 (8) | 6 (8) | 10 (12)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 1 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (13) | 6 (6) | 8 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (2) | 5 (5)
Hypochloraemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (12) | 5 (6) | 9 (17)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (10) | 3 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0) | 3 (4)
Albuminuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 3 (3) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 (10) | 8 (10) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 8 (10) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (5) | 1 (2)

LIMITATIONS AND CAVEATS:
Data and results should be interpreted with caution due to limited sample size and prematurity of data resulting from early termination and incomplete enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT05461794/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT05461794/SAP_001.pdf